CLINICAL TRIAL: NCT04455360
Title: EMERALD: Can a Virtual Eye Movement Desensitisation and Reprocessing Intervention Improve Psychological Outcome Following Covid-19 Related Critical Illness: A Feasibility Trial
Brief Title: Early EMDR Following Covid-19 Critical Illness: A Feasibility Trial
Acronym: Cov-EMERALD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Dorset HealthCare University NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Protocol version 1.2
Record Dates: First submitted 2020-06-26; First posted 2020-07-02 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Post Traumatic Stress Disorder; Intensive Care Psychiatric Disorder; Anxiety Disorders; Depression; Critical Care; COVID
Keywords: EMDR; Eye movement desensitisation and reprocessing
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression

STUDY DESIGN:
Masking Description: Patient reported outcomes at 6-months post-hospital discharge
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMDR R-TEP intervention (Experimental): Participants will receive a minimum of 2 and a maximum of 8 online EMDR R-TEP sessions, starting within 3-months of hospital discharge. Sessions will be delivered online by experienced, suitably trained and registered psychological practitioners.
  Interventions: Other: Eye Movement Desensitisation and Reprocessing Recent traumatic Event Protocol
- Standard care (No Intervention): Patients will receive standard post-hospital discharge care.

INTERVENTIONS:
Other: Eye Movement Desensitisation and Reprocessing Recent traumatic Event Protocol — EMDR is a form of psychotherapy treatment whereby the client verbally relates a narrative of a traumatic episode or emotionally disturbing material in brief sequential doses while simultaneously focusing on an external stimulus. The EMDR Recent-Traumatic Events protocol (R-TEP) aims to enable an individual to process memories of the event in order to reduce psychological morbidity. EMDR R-TEP should be delivered within 3-months of the onset of a traumatic event.
  Arms: EMDR R-TEP intervention

SUMMARY:
Primary objective is to evaluate the feasibility of delivering an online early Eye Movement Desensitisation Reprocessing (EMDR) Recent Traumatic Events Protocol (R-TEP) to patients who have survived Covid-19 related critical illness, within the context of a randomised controlled trial (RCT).

This will inform the design of a future RCT investigating the effectiveness of EMDR R-TEP in reducing psychological symptoms, for adult survivors of intensive care.

DETAILED DESCRIPTION:
A significant number of patients worldwide, have been admitted to intensive care suffering from Covid-19 related organ failure. Patients who survive a period of critical illness have a disproportionately high chance of suffering from significant and persistant poor psychological outcomes.

Eye-Movement Desensitisation and Reprocessing (EMDR) has reduced incidence of psychological morbidity in war veterans and victims of man-made and natural disasters. Small studies have also shown it to be effective in healthcare settings, within the Emergency department, following cancer diagnosis and implantation of cardioverter defibrillators. EMDR is validated by UK National Institute of Clinical Excellence guidance for use in treating adult onset PTSD.

Because of ongoing social distancing guidance our study programme aims to investigate whether it is feasible to treat patients with an early online Eye Movement Desensitisation Reprocessing (EMDR) intervention, delivered soon after hospital discharge and whether this intervention will improve psychological outcome for survivors of critical illness.

ELIGIBILITY:
Inclusion Criteria:

* Acute admission to Critical Care who have required mechanical ventilation for at least 24 hours
* PCR confirmed Covid-19 positive
* >18 years of age
* Capacity to provide informed consent

Exclusion Criteria:

* Acute brain injury
* Cognitive impairment
* Pre-existing psychotic diagnosis
* Not expected to survive post-hospital discharge
* Refusal to grant consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment, intervention adherence, incidence of treatment related adverse events and trial completion to final assessment timepoints | 12 months
  Feasibility will be determined by the following measures:
  1. Able to recruit >30% of eligible patients approached
  2. Complete early EMDR intervention programme in 75% or more of trial participants randomised to intervention.
  3. Protocol adherence
  4. Assignment of causality of serious events will be assessed by the chief investigator. Events attributable to trial procedures will be reviewed by trial management board, study sponsor and the research ethics committee, in order to determine ongoing feasibility.
  5. Outcome measures completed in 75% or more of trial participants

SECONDARY OUTCOMES:
Post-Traumatic stress disorder | 6 months post-hospital discharge
  The PTSD Checklist-Civilian Version (PCL-C) is a validated, standardised self-reporting questionnaire for PTSD comprising of 17 items that correspond to key PTSD symptoms
Anxiety and depression | 6 months
  Hospital Anxiety and Depression Scale (HADS) is a 14-item, self-reported measure with 7-items relating to symptoms of anxiety and 7-items relating to depression
Cognitive function | 6 months post-hospital discharge
  Montreal Cognitive Assessment (MoCA) is a validated tool, used to detect cogntive impairment
Health Related Quality of Life | 6 months post-hospital discharge
  EQ5D -5L comprises five quality-of-life dimensions; mobility, self-care, usual activities, pain/discomfort andanxiety/depression.
Health and disability | 6 months post-hospital discharge
  WHODAS 2.0 is a generic assessment tool that produces standarised disability levels and profiles
Physical activity | 6 months post-hospital discharge
  Wrist worn physical activity monitoring
Nutritional status | 6 months post-hospital discharge
  Patient generated subjective global assessment

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Grocott, MD, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (1):
- University Hospital Southampton NHS Foundation Trust, Southampton, Hamphsire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bates A, Golding H, Rushbrook S, Shapiro E, Pattison N, Baldwin DS, Grocott MPW, Cusack R. A randomised pilot feasibility study of eye movement desensitisation and reprocessing recent traumatic episode protocol, to improve psychological recovery following intensive care admission for COVID-19. J Intensive Care Soc. 2023 Aug;24(3):309-319. doi: 10.1177/17511437221136828. Epub 2022 Nov 19. PMID 37744073
- [Derived] Bates A, Rushbrook S, Shapiro E, Grocott M, Cusack R. CovEMERALD: Assessing the feasibility and preliminary effectiveness of remotely delivered Eye Movement Desensitisation and Reprocessing following Covid-19 related critical illness: A structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Nov 17;21(1):929. doi: 10.1186/s13063-020-04805-1. PMID 33203440